CLINICAL TRIAL: NCT01097343
Title: Clopidogrel Pharmacogenomics Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-2104
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2014-02

CONDITIONS: Disease Susceptibility
Keywords: Clopidogrel pharmacogenomics study; Performing genetic study looking at clopidogrel resistance
MeSH Terms: conditions — Disease Susceptibility | interventions — Clopidogrel

ARMS (2):
- 75 mg clopidogrel (Active Comparator)
  Interventions: Drug: clopidogrel 75 mg
- 150 mg clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel 150 mg

INTERVENTIONS:
Drug: clopidogrel 75 mg — 75 mg once daily
  Other Names: Plavix
  Arms: 75 mg clopidogrel
Drug: Clopidogrel 150 mg — clopidogrel 150 mg
  Other Names: Plavix
  Arms: 150 mg clopidogrel

SUMMARY:
Loss-of-function mutation of the gene encoding the CYP450 2C19 enzyme has emerged as a likely determinant of resistance to clopidogrel therapy. The primary hypothesis of the proposed research is that among patients with confirmed loss-of-function alleles of the CYP2C19 gene, increasing the maintenance clopidogrel dose from 75 to 150 mg will result in significant reduction in the rate of measured clopidogrel resistance defined by multiple measures of platelet function

DETAILED DESCRIPTION:
The first phase of the clinical trial will involve subject recruitment and informed consent for genetic testing. Because the target population is patients with stable coronary artery disease, patients will be recruited from the outpatient setting during clinic visits or at the time of outpatient cardiac catheterization. It is expected that all potential candidates will be initially screened for eligibility by their treating cardiologist. If a patient agrees to undergo formal screening, they will be approached by a member of the research team and receive a written summary of the clinical trial protocol that will be reviewed with the trial personnel. The initial informed consent will allow the patient to undergo genetic testing and baseline VerifyNow assay, and will also give the trial personnel permission to contact the patient by phone if they are found to be eligible for the interventional phase of the trial. The goal for enrollment in the genetic testing portion of this clinical trial is 200 patients.

If the genetic testing results confirm that the patient is a candidate for the interventional study, they will be contacted and asked to make an outpatient appointment to initiate the interventional study protocol. The therapeutic portion of this study will be a randomized, unblinded cross-over comparison of two clopidogrel dosing strategies. It is anticipated that all eligible patients will have continued their previous chronic clopidogrel therapy with standard dosing of 75 mg/day. Because all patients will be receiving chronic clopidogrel at the initiation of the intervention protocol, steady state levels should be present in all patients. Dose dependent inhibition of platelet aggregation can be seen two hours after a single oral dose of clopidogrel. Repeated doses of 75mg daily produce steady state inhibition between day 3 and day 7 of administration.

Patients who agree to participate in the therapeutic protocol, and who meet the eligibility criteria, will be randomized to an initial dosing strategy of 75 or 150 mg daily for a minimum of 30 days. At day 30 (+/- 5 days), patients will return for repeat platelet function testing. In a randomly selected subset of 15 patients, blood will be tested for the active metabolite of clopidogrel. At that time, there will be a crossover with those patients receiving 75 mg qD increased to 150 mg qD and those receiving 150 mg qD decreased to 75 mg qD. At day 60 (+/- 5 days), participants will again return for comprehensive platelet function testing and a second randomly selected group of patients will undergo testing for clopidogrel metabolites. Chronic clopidogrel dosing will be reduced to 75mg in all participants. Please see the attached schedule of events for a summary of the trial schedule.

ELIGIBILITY:
Inclusion Criteria:• Currently taking clopidogrel 75 mg/day and aspirin (minimum 81 mg/day) with an indication for chronic dual antiplatelet therapy (>90 days)

* No evidence of acute coronary syndrome within 30 days of enrollment, defined by elevation of Troponin I above the upper limit of normal
* Coronary atherosclerosis documented on previous coronary angiogram
* No known contraindications to combination therapy with aspirin and clopidogrel
* Prognosis for survival greater than one year based on physician's assessment
* Able to attend all scheduled visits.
* Access to phone
* Subject is a female with a negative urine or serum pregnancy test or post-menopausal for at least 1 year prior to randomization. Females of childbearing potential must be practicing adequate birth control to be eligible. It is the Investigator's responsibility for determining whether the Subject has adequate birth control for study participation

Exclusion Criteria:• Recent acute coronary syndrome (<30 days)

* Recent hospitalization or physician visit for bleeding disorder(<90 days) or history of chronic blood loss
* Recent blood transfusion (<90 days)
* Any contraindication to aspirin or clopidogrel therapy
* Acute Febrile illness at the time of enrollment
* Subject is pregnant or lactating or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rossi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients with 2C19*2 polymorphism were recruited to participate in a cross-over study comparing 75 vs. 150 mg of clopidogrel. 25 patients were randomized to start with 75 mg, and 25 patients started with 150 mg for 30 day dosing periods.
Pre-assignment Details: Cross-over study with two 30-day dosing periods. All patients were receiving chronic clopidogrel prior to enrollment after percutaneous coronary intervention.
Groups:
- 75 mg First 30 Days, Followed by 150 mg: 25 patients with the target allele were identified, and receive 75mg followed by 150 mg clopidogrel daily for two separate dosing periods of 30 days
- 150 mg First 30 Days, Followed by 75 mg: 25 patients with the target allele were identified, and received 150 mg clopidogrel followed by 75 mg clopidogrel for two daily for separate dosing periods of 30 days
Period: First Intervention- 30 Days
Arm/Group | 75 mg First 30 Days, Followed by 150 mg | 150 mg First 30 Days, Followed by 75 mg
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention- 30 Days
Arm/Group | 75 mg First 30 Days, Followed by 150 mg | 150 mg First 30 Days, Followed by 75 mg
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cross-over Study: All Study Participants
Arm/Group | Cross-over Study
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Clopidogrel Resistance, Defined by P2Y12 Reaction Units (PRU)Value >230
Description: P2Y12 Reaction Units are measured using the VerifyNow P2Y12 assay. Percent of patients with clopidogrel resistance defined by PRU value will be compared among low and high dose clopidogrel groups after 30 days of therapy.
Time Frame: Approximately 90 days
Population: All patients completed the clinical protocol.
Measure: Number; unit: Number of Patients with PRU>230
Groups:
- Cross-over Study- 75 mg Dose; Cross-over Study - 150 mg Dose: Participants received standard dose clopidogrel (75 mg) and higher dose (150 mg) for 30 days
Arm/Group | Cross-over Study- 75 mg Dose | Cross-over Study - 150 mg Dose
Number analyzed (Participants) | 50 | 50
Number of Patients with PRU>230 | 30 | 18
Statistical Analysis 1: Comparison: Cross-over Study- 75 mg Dose vs Cross-over Study - 150 mg Dose; A sample of size of 50 patients for the cross-over study was chosen because it provided 80% power to detect a decrease in the rate of high on-clopidogrel platelet reactivity (HPR, defined as >230 PRU) from 75% to 46% with high dose clopidogrel, with a two-sided alpha of 0.05; Test type: Superiority or Other; p = 0.02, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 90 days after enrollment in the dosing study.
Description: Adverse event data was collected during patient visits and with a follow-up phone call 30 days after completion of the dosing protocol.
Groups:
- 75 mg Followed by 150 mg; 150 mg Followed by 75 mg: Cross-over study
Arm/Group | 75 mg Followed by 150 mg | 150 mg Followed by 75 mg
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 75 mg Followed by 150 mg (N=25) | 150 mg Followed by 75 mg (N=25)
Major Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — GI bleeding requiring blood transfusion- this event occurred in a patient receiving the 150mg dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No